CLINICAL TRIAL: NCT07290582
Title: Phrenic Infiltration as Cryoanalgesia Adjuvant for Early Postoperative Pain Following the Nuss Procedure
Acronym: PHABULA
Status: Completed | Type: Observational
Sponsor: Papa Giovanni XXIII Hospital (Other)
Responsible Party: Principal Investigator, Stefano Mariconti, Medicine Doctor, Papa Giovanni XXIII Hospital
Other Study IDs: EPIC PHABULA
Record Dates: First submitted 2025-12-07; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Pectus Excavatum; Cryo Analgesia; Phrenic Nerve-related Diaphragmatic Impairment
Keywords: cryoanalgesia pectus phrenic
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EPIC: patients treated with preoperative Earlier Percutaneous Intercostal Cryoneurolysis, from 2 to 7 days prior of surgery and postoperative systemic analgesia protocol.
- PhICA: patients were treated with the same preoperative and postoperative protocol as EPIC, but adding a Phrenic Infiltration as Cryo Adjuvant, with low concentration local anesthetic, immediately after surgery and before awakening.

SUMMARY:
The goal of this observational ambispective study is to compare the effectiveness of two pain management strategies in pediatric patients undergoing the Nuss procedure for pectus excavatum. The main questions it aims to answer are:

Does the addition of phrenic Infiltration as Cryo Adjuvant (PhICA) to earlier percutaneous intercostal cryoanalgesia (EPIC) reduce postoperative pain scores compared to EPIC alone? Does the combined EPIC + PhICA technique reduce the need for rescue tramadol compared to EPIC alone? Do the two approaches differ in: length of hospital stay, time to transition to oral therapy, and time to mobilization? Are there any side effects

Researchers will compare patients who received EPIC alone to patients who received EPIC + PhICA to see if the combined technique provides superior pain control.

Participants:

Received either EPIC alone or EPIC combined with PhICA as part of their surgical anesthesia plan Had pain levels assessed using the Numeric Rating Scale (NRS) at regular postoperative intervals Were monitored for rescue tramadol requirements, medicaments taken, length of hospital stay, and mobilization timing Were monitored for any technique-related complication

DETAILED DESCRIPTION:
This is a retrospective-prospective (ambispective) study as it compares a control group (EPIC) retrospectively reviewed with a prospectively recruited case group of patients (PhICA)

ELIGIBILITY:
Inclusion Criteria:

* patients who undergo minimally invasive repair at the pediatric surgery department of our referral tertiary center

Exclusion Criteria:

* patients who refuse OR whose parents refuse to participate in the study

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adolescents and young adults with pectus excavatum undergoing the Nuss procedure for its correction
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | From surgery (Day 0) through hospital discharge, up to 7 days postoperatively.
  NRS scores of patients collected in the medical charts after surgery AND opioids consumption. For each patient, the median and the maximum pain score for each period of the day [morning (5:01-13:00) afternoon (13:01-21:00) and night (21:01-05:00)] will be computed and used as pain descriptors for statistical analyses. Opioids will be translated in morphine equivalents through validated tables.

SECONDARY OUTCOMES:
Time to mobilization after surgery | From surgery (Day 0) through hospital discharge, up to 7 days postoperatively.
  We are going to record for analysis the postoperative day (POD) in which all the following activities of daily living items were simultaneously achieved: ambulating, feeding, and toileting.
Length of hospital stay | From surgery (Day 0) through hospital discharge, up to 7 days postoperatively.
  measuring the length of hospital stay by days

OTHER OUTCOMES:
Early Anesthetic related Complications | postoperatively, From awakening up to 24 hours postoperatively, when the phrenic infiltration shows its effect before wearing off.
  Any complication related to anesthesia, particularly respiratory complications, will be assessed clinically and instrumentally (chest ultrasonography for diaphragm motion)

CONTACTS AND LOCATIONS:
Overall Officials: Ezio Bonanomi, MD, Study Chair — papa Giovanni XXIII Hospital - Bergamo
Locations (1):
- Sc Ricerca Clinica, Sviluppo E Innovazione, Bergamo, BG, Italy

IPD SHARING:
Plan to Share IPD: Undecided
We are willingful to share, as researchers, any anonymized clinical data. However, italian law is quite strict about this possibility - anyway, if requested, we will do our best to communicate.

REFERENCES:
- [Background] Hung YA, Sun CK, Chiang MH, Chen JY, Ko CC, Chen CC, Chen Y, Teng IC, Hung KC. Effect of Intraoperative Phrenic Nerve Infiltration on Postoperative Ipsilateral Shoulder Pain After Thoracic Surgeries: A Systematic Review and Meta-Analysis of Randomized Controlled Studies. J Cardiothorac Vasc Anesth. 2022 Aug;36(8 Pt B):3334-3343. doi: 10.1053/j.jvca.2022.04.016. Epub 2022 Apr 15. PMID 35570082
- [Background] Blichfeldt-Eckhardt MR, Laursen CB, Berg H, Holm JH, Hansen LN, Ording H, Andersen C, Licht PB, Toft P. A randomised, controlled, double-blind trial of ultrasound-guided phrenic nerve block to prevent shoulder pain after thoracic surgery. Anaesthesia. 2016 Dec;71(12):1441-1448. doi: 10.1111/anae.13621. Epub 2016 Sep 16. PMID 27634451
- [Result] Mariconti S, Bronco A, Pellicioli I, Chiudinelli L, Cattaneo M, Cheli M, Bonanomi E. Earlier preoperative percutaneous intercostal cryoanalgesia improves recovery after pectus excavatum surgery. Reg Anesth Pain Med. 2024 Nov 7:rapm-2024-105960. doi: 10.1136/rapm-2024-105960. Online ahead of print. PMID 39510802